CLINICAL TRIAL: NCT04837911
Title: Use of a Portable Spirometer in Pediatric Patients With Cystic Fibrosis at the Nancy CHRU: Feasibility Study
Acronym: SPIROMUCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHRU de Nancy
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis in Children

STUDY DESIGN:
Intervention Model Description: The spirometers have been purchased with charitable donations, that's why we have 35 of them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients using the Spirobank Smart (Other): Use of a portable spirometry
  Interventions: Device: Spirobank Smart

INTERVENTIONS:
Device: Spirobank Smart — Patients using the Spirobank Smart

SUMMARY:
Respiratory diseases (asthma, cystic fibrosis, COPD…) need for the diagnosis and the follow-up the use of pulmonary function tests. These technics which are used since the nineteenth century and their discovery by Hutchinson, are now currently performed in pediatrics hospitals but they require trained personnel. Spirometry can be a difficult technic, especially for children. The accuracy and repeatability depend on many factors: equipment, patient effort, supervision and encouragement of a technician. A longitudinal follow up of measures can be good especially in pediatric populations, where children have generally more difficulties recognising their symptoms.

Cystic fibrosis is a severe genetic chronic disease, that affects 1/4500 birth in France.

It's a multi system disease that affects the respiratory system, with a decline in lung function over the time and consecutive to pulmonary exacerbations, the digestive system (malabsorption of fat and vitamins) and the endocrine system (diabetes).

Pulmonary function is an important clinical indicator of the health of individuals with cystic fibrosis.

Close monitoring of patient health with daily recording of physical measurements and symptoms didn't have a negative impact, home spirometry function test could help detect earlier a decline of the lung function and pulmonary exacerbations.

Frequent exacerbations are associated with morbidity, mortality, accelerated decline in lung function and a decreased quality of life. They are also a major driver of health costs.Their early detection is a goal.

Children with cystic fibrosis have more difficulties recognizing symptoms of exacerbations.

Few studies in pediatric showed a good observance in realizing home spirometry, especially in young patients and those living far from the hospital and with a good satisfaction.

Daily monitoring of lung function is probably too tedious for children who already have lots of medication.

Medical adhesion of adolescent's patients is often suboptimal, compared with younger patients. But it's during this period that the decline of the respiratory function is the most important, with its principal cause: pulmonary exacerbations. Frequent home pulmonary function test is possible and can improve medication adherence without adding too much time, but there was no change in the decline of the FEV1 and the number of pulmonary exacerbations.

The association of home monitoring of lung function and a symptom questionary (cough, sputum and dyspnea) can predict exacerbation with a good specificity and sensibility.

The Mir Spirobank Smart is a bluetooth connected device, permitting patients to realize spirometry at home with a smartphone.

The accuracy of the Spirobank Smart compared with a spirometry in a hospital showed a good correlation (asthma and COPD population), if it's used by trained personnel.

The aim of this study is to determine the feasibility of a home respiratory monitoring in a pediatric cohort of patients with cystic fibrosis and the satisfaction of the kids, the parents and the team of the CRCM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cystic fibrosis diagnosis confirmed by a sweat chloride measurement ≥ 60 mmol/L
* Age between 10 and 20 years at enrolment
* Able to perform spirometry
* Having a smartphone
* Written consent adapted to the age
* Affiliated with a social insurance

Exclusion Criteria:

* Antibiotic therapy for a pulmonary exacerbation in the 2 weeks before enrollment
* Lung transplantation (past or future)
* Colonization with Bulkholderia cepacia in the last 2 years
* Absence of contentment
* Inability to access technology required to transmit home spirometry data
* Inability to speak and read French well enough to understand the use of the home spirometry and to complete the questionaries

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The observance of the realization of a follow up of pulmonary function in a cohort of cystic fibrosis's pediatric patients | 3 months
  Observance = the percentage (%) of measures realised during the 3 months, (number of measures done/ number of measures expected to be done according to the protocol)

SECONDARY OUTCOMES:
The workload of managing the alerts | 3 months
  The number of alerts received by each doctor and the number and therapeutic's changes following these alerts

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Mrs TATOPOULOS, Doctor, Principal Investigator — CHRU Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kruizinga MD, Essers E, Stuurman FE, Zhuparris A, van Eik N, Janssens HM, Groothuis I, Sprij AJ, Nuijsink M, Cohen AF, Driessen GJA. Technical validity and usability of a novel smartphone-connected spirometry device for pediatric patients with asthma and cystic fibrosis. Pediatr Pulmonol. 2020 Sep;55(9):2463-2470. doi: 10.1002/ppul.24932. Epub 2020 Jul 8. PMID 32592537
- [Background] Shakkottai A, Nasr SZ. The Use of Home Spirometry in Pediatric Cystic Fibrosis Patients: Results of a Feasibility Study. Glob Pediatr Health. 2017 Feb 2;4:2333794X17690315. doi: 10.1177/2333794X17690315. eCollection 2017. PMID 28229102
- [Background] Finkelstein SM, Wielinski CL, Kujawa SJ, Loewenson R, Warwick WJ. The impact of home monitoring and daily diary recording on patient status in cystic fibrosis. Pediatr Pulmonol. 1992 Jan;12(1):3-10. doi: 10.1002/ppul.1950120104. PMID 1579374
- [Background] Sarfaraz S, Sund Z, Jarad N. Real-time, once-daily monitoring of symptoms and FEV in cystic fibrosis patients--a feasibility study using a novel device. Clin Respir J. 2010 Apr;4(2):74-82. doi: 10.1111/j.1752-699X.2009.00147.x. PMID 20565480
- [Background] Shakkottai A, Kaciroti N, Kasmikha L, Nasr SZ. Impact of home spirometry on medication adherence among adolescents with cystic fibrosis. Pediatr Pulmonol. 2018 Apr;53(4):431-436. doi: 10.1002/ppul.23950. Epub 2018 Feb 19. PMID 29457700
- [Background] van Horck M, Winkens B, Wesseling G, van Vliet D, van de Kant K, Vaassen S, de Winter-de Groot K, de Vreede I, Jobsis Q, Dompeling E. Early detection of pulmonary exacerbations in children with Cystic Fibrosis by electronic home monitoring of symptoms and lung function. Sci Rep. 2017 Sep 27;7(1):12350. doi: 10.1038/s41598-017-10945-3. PMID 28955051
- [Background] Degryse J, Buffels J, Van Dijck Y, Decramer M, Nemery B. Accuracy of office spirometry performed by trained primary-care physicians using the MIR Spirobank hand-held spirometer. Respiration. 2012;83(6):543-52. doi: 10.1159/000334907. Epub 2012 Jan 21. PMID 22269344